CLINICAL TRIAL: NCT05918848
Title: Performance and Safety of Vaginal Administration of Tocopherol Acetate (Vitamin E) in Pre- Peri and Postmenopausal Women
Brief Title: Tocopherol Acetate Vaginal Administration in Pre-peri and Postmenopausal Women
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Gemelli Molise Hospital (Other)
Collaborators: Opera CRO, a TIGERMED Group Company (Other)
Responsible Party: Sponsor
Other Study IDs: GEMMOL GYNE 01/2023
Record Dates: First submitted 2023-05-11; First posted 2023-06-26 (Actual); Last update posted 2023-06-26 (Actual); Status verified 2023-06

CONDITIONS: Pre- Peri, and Postmenopausal Women
Keywords: Premenopause; perimenopause; postmenopause; vaginal eubiosis; lactobacilli flora; microbiota

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — vaginal swabs for 24 women. molecular microbiological examination for evaluation of the microbiota. The swabs were stored at -80°C to be subjected to molecular analysis
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Filme Gyno-V® Vaginal Ovules — Administration of tocopherol (Filme Gyno-V® Vaginal Ovules) for 14 days

SUMMARY:
The purpose of this non-controlled Investigator Initiated Trail (IIT), with a retrospective design is to evaluate the performance and safety of the vaginal administration of tocopherol acetate (vitamin E) in pre-peri and postmenopausal women. The main objectives of the study will be the evaluation of the vaginal pH, of the vaginal eubiosis improving the lactobacilli flora and microbiota, and of sign and symptoms of women. The patients were visited at baseline (with the collection of vaginal swabs) and treated with vaginal administration of tocopherol acetate for 14 days. At the end of treatment (final visit) the patients were visited with the collection of vaginal swabs.

DETAILED DESCRIPTION:
The vaginal microbiota has a significant bearing on a woman's mental and physical health at every stage of life. A balanced microflora of the vaginal environment (eubiosis) consists of a predominant presence of lactic acid bacteria. Lactobacilli ensure the maintenance of an acidic pH that effectively makes the environment inhospitable to pathogens by preventing infection and protecting the genital tract. At the end of the reproductive period, the reduction of sex hormones, particularly estrogen, results in a decrease in the lactobacillus component with consequent depletion of the vaginal microbiota and increased susceptibility to pathogens. Tocopherol (vitamin E) is an essential human nutrient found mainly in oily fruits. It is a fat-soluble molecule with high antioxidant power. Topically administered, it not only plays a key role in protecting epithelial cell membranes from oxidative damage but is also able to modulate bacterial growth by contributing to pH acidification. The latter feature, in the vaginal canal, creates a favorable environment for the lactobacilli flora, positively affecting the microbial population and thus contributing to the prevention of all those problems related to increased vaginal sensitivity to pathogens during "menopause." In addition, recent data show that vitamin E can counteract the production of biofilm produced by certain pathogens, which has detrimental effects on the homeostasis of the vaginal environment.

The period of observation is from January 1st, 2020 to December, 31st, 2022, while the Data Collection period will be from June, 30th, 2023 to July, 31st, 2023

ELIGIBILITY:
Inclusion Criteria:

* Women aged ≥ 50 to ≤ 70 years included.
* Premenopause, perimenopause,postmenopause women (according to STRAW criteria)
* Patients able to comply with the requirements for the study and freely willing to provide written informed consent to the retrospectively collection of their data.

Exclusion Criteria:

* Malignancy (also leukemic infiltrates) within 5 years prior to day 0 (except for treated basal cell/squamous cell carcinoma of the skin).
* Genital bleeding.
* Oestrogen topical (vaginal) treatment during the study period (it must have been terminated at least 6 months before the beginning of the study).
* Systemic oestrogen therapy during the study period (it must have been terminated at least 6 months before the beginning of the study).
* Patients with any illness, or any other medical condition, that, in the opinion of the Investigator, would compromise the participation or be likely to lead to hospitalisation during the study.
* Clinical evidence of acute infection currently requiring treatment (syphilis, herpes simplex, human papilloma virus, gonorrhoea, chlamydia, lymphogranuloma venereum, etc.); clinical evidence or history of chronic infectious disease (e.g., tuberculosis).
* Psychosis, schizophrenia, mania, depressive disorders, history of suicide attempt or suicidal ideation, or any other psychiatric illness (except for intermittent anxiety).
* Known allergy to tested medical device (tocopherol day 0.
* Participation in an interventional clinical study or administration of any investigational agents in the 30 days prior to day 0.
* Presence of any clinically significant medical condition judged by the Investigator to preclude the patient's inclusion in the study.

Ages: 50 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — The patients admitted in the Center for gynecologic visits in the period from January 1st, 2020 to December, 31st, 2022 and found eligible for inclusion in the study.
Study Population: The patients admitted in the Center for gynecologic visits in the period from January 1st, 2020 to December, 31st, 2022 and found eligible for inclusion in the study.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-06-30 (Estimated); Primary Completion 2023-07-30 (Estimated); Study Completion 2023-07-30 (Estimated)

PRIMARY OUTCOMES:
Acidity measure of vaginal secretions | 14 days
  It is assessed by Investigator during the medical examination using a pH strip (Merck, Darmstadt, Germany) with a range of 4.0 (acidic) to 7.0 (alkaline). The strip is placed on the lateral walls of the vagina to avoid contact with alkaline cervical secretions. The Investigator dip the pH test strip in the vaginal secretion for two seconds. The more acidic the vaginal secretion, the more red the strip turns, and the more alkaline the vaginal secretion, the more blue the strip turns. This provides a semiquantitative measure of pH by visually comparing the four reaction zones on the test strip to the areas of the colour scale. pH measurement serves as an indicator of the vaginal environment and the balance of microorganisms present.

SECONDARY OUTCOMES:
Rate of vaginal mucosa dryness | 14 days
  Change from baseline to 14 days assessed by the Investigator during the medical examination using a 10 cm visual analogue scale (VAS) where 0 is no dryness, and 10 is the maximum dryness.
Rate of vaginal mucosal integrity | 14 days
  Change from baseline to 14 days assessed by the Investigator during the medical examination and scored by an ordinal scale as follows: 0 = normal, 1 = superficial bleeding after scraping, 2 = superficial bleeding with light touching and 3 = presence of petechiae bleeding with light touching
Rate of mucosa pallor | 14 days
  Change from baseline to 14 days assessed by the Investigator during the medical examination and scored by a ordinal scale as follows: 0 = no pallor, 1 = slight pallor, 2 = moderate pallor, and 3 = pallor of severe intensity
Quantity of vaginal discharge assessment | 14 days
  Change from baseline to 14 days assessed by the Investigator during the medical examination and scored by a ordinal scale as follows: 0 =normal discharge overall vaginal walls, 1 = discharge covering of the vaginal walls, 2 = Scanty discharge that do not cover the entire vaginal walls, and 3 = no vaginal discharge
Whiff test | 14 days
  Change from baseline to 14 days evaluated by the following procedure: after medical examination, a sample of the vaginal discharge is placed on a glass slide, and a drop of 10% potassium hydroxide (10%KOH) is added to evaluate the presence of a fishy odour caused by the release of amine. A positive Whiff test occurs when an unpleasant odour is detected after applying the KOH solution, indicating the presence of amines. A negative Whiff test suggests the absence of this characteristic odour.
Rate of Lactobacillus grade according to Ison Hay's classification by bacterioscopic smear | 14 days
  Change from baseline to 14 days of the grade according to the modified Ison-Hay scoring system: grade 0, epithelial cells with no bacteria; grade 1, normal vaginal flora (lactobacillus morphotypes alone); grade II, reduced numbers of lactobacillus morphotypes with mixed bacterial flora; grade III, mixed bacterial flora only, few or absent lactobacillus morphotypes; grade IV, Gram-positive cocci only.
Microbiological evaluation by culture examination of the vaginal swab | 14 days
  Change from baseline to 14 days evaluated by the following procedure: the Investigator takes samples of mucus and cells from the endocervix by a swab. The samples are placed in a culture dish for a processing time of 48-72 hours to identify the presence of specific microorganisms.
Molecular sequencing-based microbiological analysis of vaginal microbiota by next-generation sequencing (NGS) method. | 14 days
  The following procedure evaluates change from baseline to 14 days: the swab is rotated in the vagina and transferred immediately on dry ice; after the sample is collected and preserved in a Copan FLOQ Sampling tube (Copan Diagnostics, Murrieta, CA, USA) at - 80 °C; the extracted DNAs are stored at - 80 °C; the sequencing is performed through the Shotgun sequencing approach. The libraries are prepared using the Illumina DNA Prep kit. The sequencing is conducted through the Illumina Novaseq 6000 system based on 2 x 150 bp paired-end reads.
  the raw reads across the samples sequences are used as input for the data analysis and finally to compare the microbiota of studied patients' groups.
Serious Adverse Device Effects / Serious Adverse Events /Adverse Device Effects/ Adverse Events | 14 days
  The number of participants with treatment-related adverse events will be assessed by CTCAE v6.0

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Cosentino, PhD, Principal Investigator — U.O.C. Ginecologia Oncologica Gemelli Molise; Roberto Di Marco, PhD, Principal Investigator — Microbiologia e Microbiologia Clinica Dipartimento Medicina e Scienze per la salute "V. Tiberio" Università degli Studi del Molise Campobasso (Italy) Laboratory

REFERENCES:
- [Background] Costantino D, Guaraldi C. Effectiveness and safety of vaginal suppositories for the treatment of the vaginal atrophy in postmenopausal women: an open, non-controlled clinical trial. Eur Rev Med Pharmacol Sci. 2008 Nov-Dec;12(6):411-6. PMID 19146203
- [Background] Palma F, Volpe A, Villa P, Cagnacci A; Writing group of AGATA study. Vaginal atrophy of women in postmenopause. Results from a multicentric observational study: The AGATA study. Maturitas. 2016 Jan;83:40-4. doi: 10.1016/j.maturitas.2015.09.001. Epub 2015 Sep 14. PMID 26421474
- [Background] Dimery IW, Hong WK, Lee JJ, Guillory-Perez C, Pham F, Fritsche HA Jr, Lippman SM. Phase I trial of alpha-tocopherol effects on 13-cis-retinoic acid toxicity. Ann Oncol. 1997 Jan;8(1):85-9. doi: 10.1023/a:1008209525671. PMID 9093712
- [Background] Panin G, Strumia R, Ursini F. Topical alpha-tocopherol acetate in the bulk phase: eight years of experience in skin treatment. Ann N Y Acad Sci. 2004 Dec;1031:443-7. doi: 10.1196/annals.1331.069. PMID 15753192
- [Background] Burton GW, Ingold KU. Vitamin E as an in vitro and in vivo antioxidant. Ann N Y Acad Sci. 1989;570:7-22. doi: 10.1111/j.1749-6632.1989.tb14904.x. PMID 2698111